CLINICAL TRIAL: NCT06638216
Title: Prospective Evaluation of Frailty in Patients With Head and Neck Tumors Before Curative Intended Therapy
Acronym: PRE-KOVERI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Prof. Dr. Franziska Hausmann, Assistant Professor for Experimental Radiation Oncology, Charite University, Berlin, Germany
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: EA1/168/24
Record Dates: First submitted 2024-10-06; First posted 2024-10-15 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Head and Neck Cancers
Keywords: Head and Neck Cancer; Frailty; Geriatric Assessment; Radiation; Maxillo-facial Surgery
MeSH Terms: conditions — Head and Neck Neoplasms; Frailty | interventions — Geriatric Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Geriatric Assessment (Experimental): Frailty is assessed using the G8 questionnaire.
  Secondary objectives include the assessment of quality of life and financial burden (EORTC-QLQ C30+ H&N43), swallowing function, cardiopulmonary resilience (6-minute walk test) and the patient's wishes regarding a prehabilitation program. Epidemiological and disease-related data is also collected.
  Interventions: Other: Geriatric Assessment

INTERVENTIONS:
Other: Geriatric Assessment — Frailty is assessed using the G8 questionnaire.
  Secondary objectives include the assessment of quality of life and financial burden (EORTC-QLQ C30+ H&N43), swallowing function, cardiopulmonary resilience (6-minute walk test) and the patient's wishes regarding a prehabilitation program. Epidemiological and disease-related data is also collected.

SUMMARY:
In a prospective study the fragility of patients with head and neck tumors before the start of curative therapy will be assessed.

Primary objective: Fragility is assessed using the G8 questionnaire.

Secondary objectives include the assessment of quality of life and financial burden (EORTC-QLQ C30+ H&N43), swallowing function, cardiopulmonary resilience (6-minute walk test) and the patient's wishes regarding a prehabilitation program. Epidemiological and disease-related data is also collected.

DETAILED DESCRIPTION:
In this prospective study patients with a tumor of the head and neck region, that are planned for Surgery or radiotherapy (chemotherapy) will be included. The probability of developing therapy-associated side effects is significantly increased if the patient is already in a limited general condition, also known as fragility, before the therapy. In addition, due to demographic change, the incidence of head and neck tumors will continue to increase, especially in patients of advanced age. Due to their age, other pre-existing conditions and infirmity, they are at a further increased risk of therapy-related side effects In order to improve the care of patients with head and neck tumors, we must first determine how many patients are affected by fragility. In addition, we want to determine influencing factors that are associated with fragility. These include, for example, difficulty swallowing and weight loss. Based on this data, we will then plan the implementation of an intervention study to establish a prehabilitation program.

ELIGIBILITY:
Inclusion Criteria:

* Indication for curative therapy in the case of an initial diagnosis of head and neck tumor disease
* Capacity to consent
* At least 18 years of age
* Sufficient knowledge of the German language

Exclusion Criteria:

* - Lack of capacity to consent
* Age <18 years
* Severe impairment of walking ability that makes it impossible to perform the 6MWT safely

Contraindications for performing a 6MWT:

Absolute contraindications* for the procedure are

* unstable angina pectoris
* myocardial infarction in the past month.

Relative contraindications are

* a resting heart rate > 120/min
* systolic blood pressure > 180 mmHg
* a diastolic blood pressure > 100 mmHg.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2024-10-07 (Actual); Primary Completion 2025-06-12 (Actual); Study Completion 2025-06-12 (Actual)

PRIMARY OUTCOMES:
Frailty | once prior to surgery or at beginning of radiation
  Assessment via G8 (Geriatric Screening Tool) questionnaire consists of 8 questions. The score ranges from 0 (poor score) to 17 points (good score), and a score of 11 or lower indicated frailty, whereas a score between 12 and 14 equals pre-frail patients. Patients with a score above 14 are considert non-frail.

SECONDARY OUTCOMES:
EORTC-QLQ C30 questionnaire | prior to surgery or at beginning of radiotherapy
  EORTC-QLQ C30 questionnaire consist of 30 questions with a score range from 0 to 100. Higher scores represents better quality of life, low scores indicating lower quality of life.
swallowing function | prior to surgery or beginning of radiation
  Questionnaire (M.D. Anderson Dysphagia Inventory), scores range from 20 (poor function) to 100 (high function)
Cardio-pulmonary resilience | prior to surgery or beginning of radiation
  6-Minute Walk test
Epidemiologic Data | prior to surgery or beginning of radiation
  Descriptive (e.g. income, alcohol use, smoking status), epidemiologic data is not scored
Information on current tumor disease | prior to surgery or beginning of radiation
  number of patients with T1/T2/T3/T4 Tumor Stage and N1/N2/N3 lymphonodal stage
EORTC-H&N43 questionnaire | prior to surgery or at beginning of radiotherapy
  EORTC-H&N43 questionnaires. Scores are from 0 to 100. A high score indicates high level of symptamotology.

CONTACTS AND LOCATIONS:
Locations (1):
- Charité University Medicine Berlin, Berlin, State of Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided